CLINICAL TRIAL: NCT03404778
Title: Comprehensive Reverse Shoulder Clinical Outcomes Study
Brief Title: Comprehensive Reverse Shoulder Data Collection
Status: Enrolling by invitation | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: ORTHO.CR.EX007
Record Dates: First submitted 2018-01-12; First posted 2018-01-19 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Arthropathy of Shoulder Region; Grossly Deficient Rotator Cuff; Osteoarthritis of the Shoulder; Rheumatoid Arthritis Without Humeral Metaphyseal Defects; Post-Traumatic Arthitis
Keywords: Reverse Shoulder Arthroplasty; Medical Device; Performance; Safety; Shoulder Prosthesis; Glenoid Erosion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Biomet Comprehensive Reverse Shoulder: Subjects in need of a reverse shoulder arthroplasty who met the inclusion/exclusion criteria and received the Comprehensive Reverse Shoulder System.
  Interventions: Device: Biomet Comprehensive Reverse Shoulder

INTERVENTIONS:
Device: Biomet Comprehensive Reverse Shoulder — Designed to eliminate the potential for scapular notching, this reverse shoulder system combines a a true locking mechanism that minimized wear and oxidative breakdown with a modular central screw for secure fixation.

SUMMARY:
This study is a multicenter, prospective, non-randomized, non-controlled clinical outcome study. The primary objective of this study is to evaluate improvement of pain score at one year for the Biomet Comprehensive Reverse Shoulder. The secondary objective is collection of long term clinical outcomes.

DETAILED DESCRIPTION:
The Biomet Comprehensive Reverse Shoulder was developed to provide an additional surgical option for patients anatomically and structurally suited to receive a reverse shoulder arthroplasty. The aim of the Biomet Comprehensive Reverse Shoulder is to increase shoulder function while reducing pain.

This is a multi-center study. Having several clinical sites will allow for multiple investigators to contribute to the results of the study. 175 implants will be included into the study. All potential study subjects will be required to participate in the Informed Consent Process.

ELIGIBILITY:
Inclusion Criteria:

* Biomet® Comprehensive™ Reverse Shoulder products are indicated for use in patients whose shoulder joint has a grossly deficient rotator cuff with severe arthropathy and/or previously failed shoulder joint replacement with a grossly deficient rotator cuff.
* The patient must be anatomically and structurally suited to receive the implants and a functional deltoid muscle is necessary.
* The Comprehensive® Reverse Shoulder is indicated for primary, fracture, or revision total shoulder replacement for the relief of pain and significant disability due to gross rotator cuff deficiency.

Exclusion Criteria:

* Absolute contraindications include infection, sepsis, and osteomyelitis.
* Uncooperative patient or patient with neurologic disorders who is incapable or unwilling to follow directions.
* Osteoporosis.
* Metabolic disorders which may impair bone formation.
* Osteomalacia.
* Distant foci of infections which may spread to the implant site.
* Rapid joint destruction, marked bone loss or bone resorption apparent on roentgenogram.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in need of a reverse shoulder arthroplasty which receive the Biomet Comprehensive Reverse Shoulder and who meet all of the inclusion and none of the exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 175 (Estimated)
Dates: Start 2010-03-07 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2036-12 (Estimated)

PRIMARY OUTCOMES:
Pain Score | 1 year
  Pain Score is assessed for each subject by asking them to indicate their current level of pain based on a 5 level scale, with "None" as the best outcome and "Severe" as the worst. Improvement of pain score at one year from pre-operative levels will be assessed.

SECONDARY OUTCOMES:
Constant Shoulder Score | Pre-operative, 3 months, 6 months, 1 year, 3 years, 5 years, 7 years, 10 years
  The Constant-Murley Shoulder Score is a scoring method used by clinicians to assess function of the shoulder. The score is on a scale of 0 to 100, with 0 being no shoulder function and 100 being excellent function.
Presence of Scapular Notching | 3 months, 6 months, 1 year, 3 years, 5 years, 7 years, 10 years
  All radiographic images collected during the study are assessed by the Principal Investigator for the presence of scapular notching. The severity of notching will be assessed using the Nerot system, where Grade 0 indicates no notch and Grade 4 indicates the largest-sized defect in the scapula.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Acromion LLC, Towson, Maryland
  - William Beaumont Hospital, Royal Oak, Michigan
  - Allina Health System DBA Sports and Orthopaedic Specialists, Edina, Minnesota
  - Joint Implant Surgeons, New Albany, Ohio